CLINICAL TRIAL: NCT06735339
Title: A New Organisation of Healthcare for Multimorbidity
Brief Title: A New Organisation of Clinic for Multimorbidity and Polypharmacy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1-16-02-342-24; 1-16-02-342-24 (Registry Identifier: Central Denmark Region's registry of research projects)
Record Dates: First submitted 2024-12-03; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Multimorbidity
Keywords: multimorbidity; continuity of care; patient pathway; Denmark; outpatient care; multidisciplinary; MDT; appropriate medicine; comorbidity
MeSH Terms: interventions — Ambulatory Care Facilities; Multimorbidity

STUDY DESIGN:
Intervention Model Description: Stepped-wedge randomised design including 6 hospital clusters of general practitioners in the Central Denmark Region.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinic for multimorbidity (Experimental): All participants will be assigned to the intervention but at different times according to the stepped wedge design. There are 6 clusters, to be assigned at different times.
  Interventions: Other: Clinic for Multimorbidity

INTERVENTIONS:
Other: Clinic for Multimorbidity — The patient is assigned a healthcare coordinator. A review of the patient's medication history and a medication review are conducted. A functional assessment is performed, along with relevant measurements, and the patient consults with a specialist physician. A multidisciplinary team (MDT) conference is held with selected specialists, depending on the patient's needs. This may include a cardiologist, endocrinologist, pulmonologist, gastroenterologist, rheumatologist, nephrologist, geriatrician, clinical pharmacologist, psychiatrist, pain nurse, physiotherapist, occupational therapist, and the patient's GP.
  The handover of information to the GP is agreed upon at the time of referral and can be carried out in writing, through virtual MDT participation, or by telephone.
  In agreement with the patient, the clinic may initiate follow-up actions, such as counseling on medication or disease management. Additionally, the clinic may facilitate cross-sectoral activities, such as therapy.

SUMMARY:
The purpose of this study is to investigate:

1) the implementation and 2) the effects of an outpatient program for patients with complex multimorbidity. The investigators intend to integrate care from various health professionals across medical specialties and sectors, promote person-centered care, and ensure a holistic approach. Specifically, the investigators have redesigned the existing clinic, the Clinic for Multimorbidity, which has been operational since 2012 without any protocol-based evaluation. The new version introduces differentiated care options based on general practitioners needs for support.

Multimorbidity, defined as the presence of two or more chronic diseases in an individual, poses a significant challenge for healthcare systems globally. There is an urgent need for targeted interventions for those with high complexity, such as due to interacting diseases and polypharmacy, particularly in light of an aging population, where on-fourth has multimorbid. Although the care for individuals with multimorbidity often may be perceived as fragmented, there is limited evidence on how to best organize the care. Effective, evidence-based strategies to ensure integration are lacking.

The population will consist of adults with complex multimorbidity from the Central Denmark Region, referred to the Clinic for Multimorbidity from general practice. Using a stepped wedge randomized controlled design, the project will encompass two studies.

1. The implementation study will be based on implementation outcomes by Proctor et al: acceptability, adoption, appropriateness, feasibility, fidelity, and penetration. Data will be collected through interviews with patients and general practitioners, as well as measurements related to referral practices, costs, and feasibility.
2. The effectiveness study will include outcome measures such as questionnaire-based patient experiences regarding health-related quality of life, treatment burden, depression, and anxiety. Additionally, the investigators will assess effects on inappropriate medication, symptoms, mortality, treatment continuity, healthcare utilization, and the initiation of health-promoting initiatives.

The investigators anticipate demonstrating that multimorbid patients will benefit from an interdisciplinary, cross-sector collaborative model. Furthermore, the investigators expect that this new organization will support general practitioners, municipalities, and hospitals in their management of these patients, addressing differentiated treatment needs in accordance with the recommendations of the Danish Health Structure Commission.

ELIGIBILITY:
Inclusion Criteria:

* Aged18 years or older
* Multimorbidity: = 2 chronic conditions (minimum 6 months' duration per condition)
* Polypharmacy (= 5 medications)
* Complexity: Complex multimorbidity refers to the patient suffering from multiple concurrent, chronic diseases/conditions creating additional challenges. Complexity can be of physical, mental, social character and due to medication, high treatment burden, frailty, frequent healthcare visits or a special need for joint healthcare collaboration.

Exclusion criteria:

Diagnostically unresolved conditions and patients whose primary issues require focused management of chronic pain, psychiatric disorders, alcohol misuse, and other addiction-related challenges.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-05 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Need-based quality of life (MMQ-1 questionnaire) | From enrollment to 3 months after have undergone a trajectory at Clinic for Multimorbidity
  Will be assessed using the MultiMorbidity Questionnaire MMQ-1 measuring needs-based QoL: physical ability (6 items), worries (6 items), limitations in everyday life (10 items), social life (6 items), self-image (6 items), and personal finances (3 items). -in total 31 items.
  The questionnaire was deveoped by Bissenbakker et al. and has been validated in Danish settings for patients living with multimorbidity: the MMQ1 is a condition-specific PROM with adequate psychometric properties designed to measure needs-based QoL.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for Multimorbidity, Medical Diagnostic Centre, Central Denmark Region, Denmark, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://ijic.org/articles/10.5334/ijic.7015